CLINICAL TRIAL: NCT01100385
Title: Vascular Effects of Nutritional Supplementation With a Standardised Preparation of Tomato Extract (Ateronon) in Vivo in Man
Brief Title: TomVasc - Vascular Effects of Tomato Extract
Acronym: TomVasc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: Cambridge Theranostics Ltd (Industry)
Responsible Party: Principal Investigator, Joseph Cheriyan, MD, Consultant Physician, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: A091763; 09/H03011/106 (Other: REC)
Record Dates: First submitted 2010-04-08; First posted 2010-04-09 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2012-07

CONDITIONS: Ischemic Heart Disease; Transient Ischemic Attack; Stroke; Peripheral Vascular Disease
Keywords: Healthy adults
MeSH Terms: conditions — Myocardial Ischemia; Ischemic Attack, Transient; Stroke; Peripheral Vascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Healthy (placebo) (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Healthy (Ateronon) (Active Comparator)
  Interventions: Dietary Supplement: Ateronon
- Cardiovascular Group (placebo) (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Cardiovascular Group (Ateronon) (Active Comparator)
  Interventions: Dietary Supplement: Ateronon

INTERVENTIONS:
Dietary Supplement: Ateronon — Tomato extract (lycopene) capsule, taken once daily for 56 days
  Arms: Cardiovascular Group (Ateronon); Healthy (Ateronon)
Dietary Supplement: Placebo — Matched placebo capsule, taken once daily for 56 days
  Arms: Cardiovascular Group (placebo); Healthy (placebo)

SUMMARY:
Does tomato extract improve blood vessel function in healthy people and people with cardiovascular disease?

Atherosclerosis ('furring' of the arteries) affects the functioning of blood vessels, narrowing and eventually blocking them, causing conditions like heart attack and stroke. The Mediterranean diet, which is rich in tomatoes and tomato-based products, has been shown to be associated with a reduced risk of blood vessel damage. In this double blind, placebo-controlled randomised study, the investigators will investigate whether a food supplement containing a standardised extract of tomato improves blood vessel function in both healthy people (aged 40-80), and people with a history of cardiovascular disease. The food supplement is on sale to the public, and the investigators are testing the standard dose. Approximately 72 people will take part at the Clinical Pharmacology Unit at the ACCI Building, Cambridge University Hospitals NHS Trust.

After they have passed screening tests, participants will be allocated by chance to receive either the tomato extract product (Ateronon), or a matching placebo (a dummy capsule with no active ingredients), which they will take once a day for 8 weeks. At the beginning and end of the treatment period, the investigators will test blood vessel stiffness using an ECG machine and external probe. The investigators will also measure forearm blood flow, which involves infusing 3 separate agents that affect how the lining of the blood vessel wall works, and helps to assess whether this is affected by the study treatment. Blood tests will also be used to look at how the food supplement is working and its effects on cholesterol and markers of inflammation. Including the screening period, and a follow-up telephone call two weeks after the end of treatment, participants will be in the study for 14 weeks.

ELIGIBILITY:
HEALTHY GROUP

Inclusion Criteria:

* Aged between 30 and 80 years
* Non-smoking

Exclusion Criteria:

* Hypertension or other cardiovascular disease
* Significant renal, respiratory or neurological disease
* Diabetes mellitus
* BMI>32, BMI<18
* Use of vasoactive medication
* Use of heparin or warfarin
* Allergy/intolerance to study substance ingredients

STABLE CARDIOVASCULAR DISEASE GROUP

Inclusion Criteria:

* Aged between 40 and 80 years
* Previous ischaemic heart disease (any of previous myocardial infarction, coronary stent, angina), transient ischaemic attack or stroke disease or peripheral vascular disease
* If taking a statin, dose must have been stable over preceding 2 months

Exclusion Criteria:

* Uncontrolled hypertension
* BMI>33
* Use of heparin or warfarin
* Allergy/intolerance to study substance ingredients

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2010-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Forearm blood flow ratio and/or absolute flow in the infused arm (and % change), as measured by venous occlusion plethysmography, in response to intra-arterial acetylcholine infusion. | 8 weeks

SECONDARY OUTCOMES:
Forearm blood flow ratio and/or absolute flow in the infused arm (& % change), as measured by venous occlusion plethysmography, in response to intra-arterial sodium nitroprusside and L-NMMA infusion. | 8 weeks
Evaluation of pulse wave velocity and pulse wave analysis | 8 weeks
Pulse wave velocity measured between carotid and femoral artery. | 8 weeks
Analysis of Lipoprotein oxidation/circulating markers. | 8 weeks
Safety and tolerability parameters, including physical examination, blood pressure, heart rate, 12-lead electrocardiograms (ECGs), clinical laboratory tests and adverse event reporting. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dr Joseph Cheriyan, MBChB, MRCP, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Addenbrooke's Hospital, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- [Derived] Gajendragadkar PR, Hubsch A, Maki-Petaja KM, Serg M, Wilkinson IB, Cheriyan J. Effects of oral lycopene supplementation on vascular function in patients with cardiovascular disease and healthy volunteers: a randomised controlled trial. PLoS One. 2014 Jun 9;9(6):e99070. doi: 10.1371/journal.pone.0099070. eCollection 2014. PMID 24911964